CLINICAL TRIAL: NCT02328482
Title: A Pivotal, Multicenter, Open-label, Randomized Withdrawal, Non-Treatment Concurrent Control Study to Assess the Safety, Tolerability, and Efficacy of Cabaletta® in OPMD Patients Who Participated in Study BBCO-001
Brief Title: Continuation Protocol to Protocol BBCO-001
Acronym: HOPEMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioblast Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB-OPMD-301
Record Dates: First submitted 2014-12-25; First posted 2014-12-31 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2018-02

CONDITIONS: Muscular Dystrophy, Oculopharyngeal (OPMD)
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Oculopharyngeal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Trehalose 30 g for IV infusion administered every week over an additional 52 weeks
  Interventions: Drug: Tehalose 30gr
- Arm 2 (No Intervention): no-treatment concurrent control; follow-up over 52 weeks

INTERVENTIONS:
Drug: Tehalose 30gr — Trehalose 30 g for IV infusion administered every week over an additional 52 weeks
  Other Names: Cabellta
  Arms: Arm 1

SUMMARY:
This will be a multi-center, randomized withdrawal, open-label, non-treatment concurrent control, parallel group study. Patients completing protocol BBCO-001 will be offered the opportunity to enter into this 12-month randomized withdrawal protocol.

DETAILED DESCRIPTION:
This will be a multi-center, randomized withdrawal, open-label, non-treatment concurrent control, parallel group study. Patients completing protocol BBCO-001 will be offered the opportunity to enter into this 12-month randomized withdrawal protocol.

Eligible patients will be randomized to one of the following treatment arms:

* Treatment Arm 1: active treatment; continuation of 30 g IV Cabaletta once a week over an additional 52 weeks.
* Treatment Arm 2: no-treatment concurrent control; discontinuation of IV Cabaletta and follow-up over 52 weeks.

IV Cabaletta will be administered once a week to patients in Treatment Arm 1. All patients, regardless of treatment arm allocation, will undergo the same safety and efficacy assessments during the monthly site visits.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women who participated and completed study BBCO-001
2. Clinical and genetic diagnosis of OPMD
3. Able to provide written informed consent to participate in this study
4. Able to understand the requirements of the study and willing to comply with the requirements of the study

Exclusion Criteria:

1. Pregnant or lactating
2. Currently receiving anticoagulant treatment (e.g., warfarin)
3. Any life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety
4. Known hypersensitivity to any ingredient in the Cabaletta IV infusion
5. Currently participating in another clinical trial (other than BBCO-001) or have completed an interventional trial less than 30 days prior to the planned treatment start date

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in disease markers | 52 weeks
  long term effect of Cabaletta on disease progression as measured by the changes in the disease markers
Change in swallowing quality of life | 52 weeks
  long term effect of Cabaletta on disease progression as measured by the changes in the patient's swallowing quality of life

SECONDARY OUTCOMES:
Long-term safety and tolerability of repeated intravenous (IV) of Cabaletta 30 g | 52 weeks
  The safety and tolerability will be evaluated by measuring the adverse events, vital signs, safety labs and physical examination during the entire study period. The number of events of change in the safety evaluations will be compared between the treatment and non treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Brais, Principal Investigator — McGill University
Locations (1):
- Montreal Neurological Institute, McGill University, Montreal, Quebec, Canada